CLINICAL TRIAL: NCT03372850
Title: A Randomized, Open-label, Multiple Dose, Crossover Study to Compare the Safety, Pharmacokinetics and Pharmacodynamics of HIP1601 (40 mg or 20 mg) to HGP1705 (40 mg or 20 mg) After Multiple Administrations in Healthy Male Volunteers
Brief Title: Safety, Pharmacokinetics and Pharmacodynamics of the Two Esomeprazole Formulations
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HM-ESOM-101
Record Dates: First submitted 2017-12-08; First posted 2017-12-14 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Healthy
MeSH Terms: interventions — Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence Group 1 (Experimental): Period 1: Reference Drug(HGP1705) Period 2: Test Drug(HIP1601)
  Interventions: Drug: HIP1601; Drug: HGP1705
- Sequence Group 2 (Experimental): Period 1: Test Drug(HIP1601) Period 2: Reference Drug(HGP1705)
  Interventions: Drug: HIP1601; Drug: HGP1705

INTERVENTIONS:
Drug: HIP1601 — Test Drug
  Other Names: Esomeprazole (40 mg or 20 mg)
Drug: HGP1705 — Reference Drug
  Other Names: Nexium(esomeprazole 40 mg or 20 mg)

SUMMARY:
This study is a Randomized, Open-label, Multiple Dose, Crossover Study to Compare the Safety, Pharmacokinetics and Pharmacodynamics of HIP1601 (40 mg or 20 mg) to HGP1705 (40 mg or 20 mg) After Multiple Administrations in Healthy Male Volunteers

DETAILED DESCRIPTION:
This study is a 2-part study, where in Part A, the 40 mg dose will be performed followed by the 20 mg dose in Part B.

ELIGIBILITY:
Inclusion Criteria:

1. Age 19~50 years in healthy male volunteers
2. BMI is more than 18 kg/m^2 , no more than 27.0 kg/m^2
3. Subjects who have ability to comprehend the objectives, contents of study and property of study drug before participating in trial and have willingness to sign of informed consent in writing

Exclusion Criteria:

1. Presence of medical history or a concurrent disease that may interfere with treatment and safety assessment or completion of this clinical study, including clinically significant disorders in digestive system, neuropsychiatric system, endocrine system, liver, cardiovascular system
2. Subjects who judged ineligible by the investigator

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2018-02-15 (Estimated); Primary Completion 2018-06-15 (Estimated); Study Completion 2018-06-15 (Estimated)

PRIMARY OUTCOMES:
AUClast of esomeprazole | 1 Day 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 10, 12, 16, 4 Day 0 hour, 5 Day 0 hour, 6 Day 0 hour, 7 Day 0 hour, 8 Day 0 hour
  pharmacokinetic evaluation
After 7days of repeated administration, Total gastric acidity decrease rate versus baseline for 24 hours | 7Day 24h(Full time) pH monitoring
  pharmacodynamic evaluation

SECONDARY OUTCOMES:
AUCinf of esomeprazole | 1 Day 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 10, 12, 16, 4 Day 0 hour, 5 Day 0 hour, 6 Day 0 hour, 7 Day 0 hour, 8 Day 0 hour
  pharmacokinetic evaluation
Cmax of esomeprazole | 1 Day 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 10, 12, 16, 4 Day 0 hour, 5 Day 0 hour, 6 Day 0 hour, 7 Day 0 hour, 8 Day 0 hour
  pharmacokinetic evaluation
Tmax of esomeprazole | 1 Day 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 10, 12, 16, 4 Day 0 hour, 5 Day 0 hour, 6 Day 0 hour, 7 Day 0 hour, 8 Day 0 hour
  pharmacokinetic evaluation
Terminal Half-life of esomeprazole | 1 Day 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 10, 12, 16, 4 Day 0 hour, 5 Day 0 hour, 6 Day 0 hour, 7 Day 0 hour, 8 Day 0 hour
  pharmacokinetic evaluation
CL/F of esomeprazole | 1 Day 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 10, 12, 16, 4 Day 0 hour, 5 Day 0 hour, 6 Day 0 hour, 7 Day 0 hour, 8 Day 0 hour
  pharmacokinetic evaluation
Vd/F of esomeprazole | 1 Day 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 10, 12, 16, 4 Day 0 hour, 5 Day 0 hour, 6 Day 0 hour, 7 Day 0 hour, 8 Day 0 hour
  pharmacokinetic evaluation
Ctrough | 1 Day 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 51 Day 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 10, 12, 16, 2 Day 0 hour
  pharmacokinetic evaluation
Ctrough,ss | 1 Day 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 10, 12, 16, 4 Day 0 hour, 5 Day 0 hour, 6 Day 0 hour, 7 Day 0 hour, 8 Day 0 hour
  pharmacokinetic evaluation
PTF | 1 Day 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 10, 12, 16, 4 Day 0 hour, 5 Day 0 hour, 6 Day 0 hour, 7 Day 0 hour, 8 Day 0 hour
  pharmacokinetic evaluation
RActrough | 1 Day 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 10, 12, 16, 4 Day 0 hour, 5 Day 0 hour, 6 Day 0 hour, 7 Day 0 hour, 8 Day 0 hour
  pharmacokinetic evaluation
After the first administration of esomeprazole, The rate of decrease of integrated gastric acidity compared to baseline for 24 hours | 1Day 24h pH monitoring
  pharmacodynamic evaluation
After the first dose and 7 days of repeated dosing, Percentage of time to maintain gastric pH 4.0 or higher for 24 hours | 1Day(Full time) pH monitoring, 7Day 24h(Full time) pH monitoring
  pharmacodynamic evaluation
After the first administration and 7 days of repeated administration, The median pH measured for 24 hours | 1Day(Full time) pH monitoring, 7Day 24h(Full time) pH monitoring
  pharmacodynamic evaluation
After first administration and 7 days of repeated administration, Total gastric acidity reduction rate versus baseline between 12hours and 24 hours | 1Day 12h, 2Day 0h, 7Day 12h, 8Day 0h
  pharmacodynamic evaluation
After the first dose and 7 days of repeated dosing, Percentage of time to maintain gastric pH 4.0 or higher between 12hours and 24 hours | 1Day 12h, 2Day 0h, 7Day 12h, 8Day 0h
  pharmacodynamic evaluation
After the first dose and 7 days of repeated dosing, The median pH measured between 12hours and 24 hours | 1Day (12~24h) pH monitoring, 7Day (12~24h) pH monitoring
  pharmacodynamic evaluation

OTHER OUTCOMES:
After first administration and repeated administration for 7 days, The percentage of decrease in integrated gastric acidity compared to baseline by time | 1Day(Full time) pH monitoring, 7Day 24h (Full time) pH monitoring
  exploratory endpoint

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No